CLINICAL TRIAL: NCT01415882
Title: Phase 2 Trial of Ixazomib Combinations in Patients With Relapsed Multiple Myeloma
Brief Title: Ixazomib Citrate in Treating Patients With Relapsed Multiple Myeloma That Is Not Refractory to Bortezomib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1181; NCI-2011-02303 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-001516 (Other: Mayo Clinic Institutional Review Board); MC1181 (Other: Mayo Clinic)
Record Dates: First submitted 2011-08-05; First posted 2011-08-12 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (ixazomib citrate and dexamethasone, closed to accrual) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15. Patients with lack of minor response by the end of the second cycle or lack of partial response by the end of the fourth cycle also receive dexamethasone PO on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis
- Arm B (ixazomib citrate and dexamethasone) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15 and dexamethasone PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis
- Arm C (higher-dose ixazomib citrate and dexamethasone) (Experimental): Patients receive higher doses of ixazomib citrate PO on days 1, 8, and 15 and dexamethasone PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis
- Arm D (ixazomib citrate, dexamethasone, and cyclophosphamide) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO (cycles 1-18 only) and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis
- Arm E (ixazomib citrate, cyclophosphamide, daratumumab) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15, cyclophosphamide PO (cycles 1-12 only) on days 1, 8, 15, 22, and daratumumab IV on days 1, 8, 15, 22 (cycles 1-2), days 1 and 15 (cycles 3-6), and day 1 in all subsequent cycles. Patients also receive dexamethasone IV or PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Daratumumab; Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm D (ixazomib citrate, dexamethasone, and cyclophosphamide); Arm E (ixazomib citrate, cyclophosphamide, daratumumab)
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
  Arms: Arm E (ixazomib citrate, cyclophosphamide, daratumumab)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ixazomib citrate works in treating patients with multiple myeloma that has returned after a period of improvement (relapsed) but is not resistant to bortezomib (refractory). Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the confirmed overall response rate (>= partial response [PR]) of ixazomib [ixazomib citrate], used as a single agent in patients with relapsed multiple myeloma, who are proteasome inhibitor naive (including bortezomib) naive OR have received less than 6 cycles of therapy with bortezomib and had a better than PR with no progression at the time of discontinuation. (Arm A - Permanently closed to accrual as of Addendum 5) II. To determine the confirmed overall response rate (>= PR) of ixazomib at a 4 mg dose level in combination with dexamethasone in patients with relapsed multiple myeloma, who are proteasome inhibitor naive (including bortezomib) naive OR have received less than 6 cycles of therapy with bortezomib and had a better than PR with no progression at the time of discontinuation. (Arm B) III. To determine the confirmed overall response rate (>= PR) of ixazomib at a 5.5 mg dose level in combination with dexamethasone in patients with relapsed multiple myeloma, who are proteasome inhibitor naive (including bortezomib) naive OR have received less than 6 cycles of therapy with bortezomib and had a better than PR with no progression at the time of discontinuation. (Arm C) IV. To determine the confirmed overall response rate (>= PR) of ixazomib in combination with cyclophosphamide and dexamethasone in patients with relapsed multiple myeloma, who are proteasome inhibitor naive (including bortezomib) naive OR have received less than 6 cycles of therapy with bortezomib and had a better than PR with no progression at the time of discontinuation. (Arm D) V. To determine the confirmed overall response rate (>= PR) of ixazomib in combination with cyclophosphamide, daratumumab, and dexamethasone in patients with relapsed multiple myeloma. (Arm E)

SECONDARY OBJECTIVES:

I. To determine the overall response rate of ixazomib in combination with dexamethasone, when dexamethasone is added to ixazomib for lack of response or for progression. (Arm A) II. To determine the event free survival and overall survival among patients with relapsed myeloma following treatment with ixazomib with dexamethasone added for lack of response or progression. (Arm A) III. To determine the event free survival and overall survival among patients with relapsed myeloma following treatment with ixazomib at two different doses, in combination with dexamethasone. (Arms B and C) IV. To determine the event free survival and overall survival among patients with relapsed myeloma following treatment with ixazomib in combination with cyclophosphamide and dexamethasone. (Arm D) V. To determine the event free survival and overall survival among patients with relapsed myeloma following treatment with ixazomib in combination with cyclophosphamide, daratumumab, and dexamethasone. (Arm E)

OUTLINE: Patients are randomized to 1 of 4 treatment arms (Arm A permanently closed to accrual as of Addendum 5).

ARM A: Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15. Patients with lack of minor response by the end of the second cycle or lack of partial response by the end of the fourth cycle also receive dexamethasone PO on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive ixazomib citrate PO on days 1, 8, and 15 and dexamethasone PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive higher dose of ixazomib citrate PO on days 1, 8, and 15 and dexamethasone PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO (cycles 1-18 only) and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive ixazomib citrate PO on days 1, 8, and 15, cyclophosphamide PO (cycles 1-12 only) on days 1, 8, 15, 22, and daratumumab intravenously (IV) on days 1, 8, 15, 22 (cycles 1-2), days 1 and 15 (cycles 3-6), and day 1 in all subsequent cycles. Patients also receive dexamethasone IV or PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 or 12 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min (obtained =< 14 days prior to registration)
* Absolute neutrophil count >= 1000/mL (obtained =< 14 days prior to registration)
* Untransfused platelet count >= 75000/mL (obtained =< 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (obtained =< 14 days prior to registration)
* Patients with relapsed multiple myeloma who have already received one or more standard treatment regimens
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * For patients with extramedullary disease (EMD) measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) or the CT portion of the positron emission tomography (PET)/CT: Must have at least one lesion that has a single diameter of >= 2 cm. Skin lesions can be used if the area is >= 2 cm in at least one diameter and measured with a ruler
  * Plasma cell count >= 0.5 x 10^9/L or 5 percent of the peripheral blood white cells
  * Plasma cell count if determined by flow cytometry, >= 200/150,000 events
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to return to consenting Mayo Clinic institution for follow-up during the Active Monitoring Phase of the study; Note: during the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Recovered (i.e., < grade 1 toxicity) from the reversible effects of prior antineoplastic therapy
* Arms A - D only: Patients should be proteasome inhibitor naive (including bortezomib and carfilzomib) OR have received less than 6 cycles of therapy with a bortezomib or carfilzomib containing regimen and were not refractory to the bortezomib or carfilzomib based regimen (less than a PR or progression on or within 60 days of discontinuation)
* Arm E only: Negative hepatitis B test (defined by a negative test for hepatitis B surface antigen [HBsAg], or antibodies to hepatitis B surface and/or core antigens [antiHBs or antiHBc]) (added as of addendum 9); Note: patients with serologic findings suggestive of hepatitis B virus (HBV) vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR); those who are PCR positive will be excluded

Exclusion Criteria:

* Recent prior chemotherapy:

  * Alkylators (e.g. melphalan, cyclophosphamide) =< 14 days prior to registration
  * Anthracyclines =< 14 days prior to registration
  * High dose corticosteroids, immune modulatory drugs (thalidomide or lenalidomide) =< 7 days prior to registration
* Prior therapy with any proteasome inhibitor other than bortezomib, carfilzomib, or ixazomib
* Concomitant high dose corticosteroids other than what is part of treatment protocol (concurrent use of corticosteroids); EXCEPTION: patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, i.e., adrenal insufficiency, rheumatoid arthritis, etc
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use 2 effective methods of contraception from the time of signing the informed consent form through 90 days after the last dose of study drug
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 30 days after stopping treatment
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Major surgery within 14 days before study registration
* Systemic treatment with strong inhibitors of cytochrome P450, family 1, subfamily A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months; Note: prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diarrhea > grade 1, based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grading, in the absence of antidiarrheals
* Arm E only: Refractory to any combination of a proteasome inhibitor and daratumumab
* Arm E only: Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. (Note that FEV1 testing is required for subjects suspected of having chronic obstructive pulmonary disease and subjects must be excluded if FEV1 < 50% of predicted normal.)
* Arm E only: Known moderate or severe persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Kumar SK, LaPlant BR, Reeder CB, Roy V, Halvorson AE, Buadi F, Gertz MA, Bergsagel PL, Dispenzieri A, Thompson MA, Crawley J, Kapoor P, Mikhael J, Stewart K, Hayman SR, Hwa YL, Gonsalves W, Witzig TE, Ailawadhi S, Dingli D, Go RS, Lin Y, Rivera CE, Rajkumar SV, Lacy MQ. Randomized phase 2 trial of ixazomib and dexamethasone in relapsed multiple myeloma not refractory to bortezomib. Blood. 2016 Nov 17;128(20):2415-2422. doi: 10.1182/blood-2016-05-717769. Epub 2016 Oct 4. PMID 27702799
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Ixazomib Citrate and Dexamethasone): Patients receive ixazomib citrate PO on days 1, 8, and 15. Patients with lack of minor response by the end of the second cycle or lack of partial response by the end of the fourth cycle also receive dexamethasone PO on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone) | Arm B (Ixazomib Citrate and Dexamethasone) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab)
Started | 33 | 36 | 35 | 37 | 24
Completed | 32 | 35 | 35 | 33 | 24
Not Completed | 1 | 1 | 0 | 4 | 0
Not completed — Ineligible | 1 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone, Closed to Accrual) | Arm B (Ixazomib Citrate and Dexamethasone) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab) | Total
Number analyzed (Participants) | 33 | 36 | 35 | 37 | 24 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.4) | 70.0 (8.4) | 67.8 (7.9) | 69.1 (10.6) | 68.1 (8.7) | 68.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 13 | 15 | 6 | 68
  Male | 18 | 17 | 22 | 22 | 18 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 1 | 0 | 6
  Not Hispanic or Latino | 30 | 34 | 32 | 36 | 24 | 156
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 33 | 36 | 35 | 36 | 24 | 164
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Confirmed Responses With Ixazomib Citrate Alone (Arm A [Closed]), Ixazomib Citrate With Dexamethasone (Arms B + C), or With Dexamethasone and Cyclophosphamide (Arm D), or With Dexamethasone, Cyclophosphamide, Daratumumab (Arm E)
Description: A confirmed response is defined as stringent complete response, complete response (CR), very good partial response, or partial response (PR) noted as the objective status on 2 separate evaluations while receiving ixazomib citrate with or without dexamethasone. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. 95% confidence intervals for the true success proportion will be calculated by the exact binomial method.
Time Frame: 2.5 years
Population: All eligible patients that received treatment and a disease evaluation.
Measure: Number; unit: proportion of participants
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone) | Arm B (Ixazomib Citrate and Dexamethasone) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab)
Number analyzed (Participants) | 32 | 35 | 35 | 36 | 24
proportion of participants | 0.1563 | 0.3143 | 0.5429 | 0.6667 | 0.750

2. Secondary Outcome: Confirmed Response Rate With the Addition of Dexamethasone (Arm A Only)
Description: Estimated by the number of patients who achieve a confirmed response at any time (with single agent ixazomib citrate or ixazomib citrate plus dexamethasone) divided by the number of evaluable patients. 95% confidence intervals for the true confirmed response rate will be calculated by the exact binomial method.
Time Frame: 2.5 years
Measure: Number; unit: proportion of participants
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone)
Number analyzed (Participants) | 32
proportion of participants | 0.3438

3. Secondary Outcome: Overall Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: 2.5 years
Population: All eligible patients that started treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone) | Arm B (Ixazomib Citrate and Dexamethasone) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab)
Number analyzed (Participants) | 32 | 35 | 35 | 33 | 24
Months | NA [NA to NA] — Not enough events occurred to calculate the Median or confidence intervals | NA [26.3 to NA] — Not enough events occurred to calculate the Median or upper confidence interval | NA [25.5 to NA] — Not enough events occurred to calculate the Median or upper confidence interval | NA [NA to NA] — Not enough events occurred to calculate the Median or confidence intervals | NA [NA to NA] — Not enough events occurred to calculate the Median or confidence intervals

4. Secondary Outcome: Event-free Survival
Description: Date of progression will be defined as the date that the criteria for progressive disease were first met after initiation of dexamethasone. The distribution of event-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to disease progression while receiving ixazomib citrate and dexamethasone, death due to any cause, or subsequent treatment for multiple myeloma, assessed up to 2.5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone) | Arm B (Ixazomib Citrate and Dexamethasone) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab)
Number analyzed (Participants) | 32 | 35 | 35 | 33 | 24
Months | 11.5 [9.1 to 20.3] | 8.4 [4.5 to 12.8] | 7.8 [4.6 to 11.9] | 18.8 [10.2 to 30.4] | 29.5 [18.8 to 39.6]

5. Secondary Outcome: Incidence of Adverse Events
Description: Graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The maximum grade for each type of adverse event, regardless of causality, will be recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Time Frame: Up to 30 days after the last day of study drug treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Arm A (Ixazomib Citrate and Dexamethasone) | Arm B (Ixazomib Citrate and Dexamethasone) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab)
All-Cause Mortality (participants affected / at risk) | 5/33 | 5/35 | 4/35 | 8/36 | 6/24
Serious Adverse Events (participants affected / at risk) | 16/33 | 11/35 | 11/35 | 14/36 | 14/24
Other Adverse Events (participants affected / at risk) | 33/33 | 35/35 | 35/35 | 36/36 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ixazomib Citrate and Dexamethasone) (N=33) | Arm B (Ixazomib Citrate and Dexamethasone) (N=35) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) (N=35) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) (N=36) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab) (N=24)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Lung infection (Infections and infestations) | 3 (4) | 4 (6) | 1 (1) | 2 (2) | 3 (5)
Sepsis (Infections and infestations) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ixazomib Citrate and Dexamethasone) (N=33) | Arm B (Ixazomib Citrate and Dexamethasone) (N=35) | Arm C (Higher-dose Ixazomib Citrate and Dexamethasone) (N=35) | Arm D (Ixazomib Citrate, Dexamethasone, and Cyclophosphamide) (N=36) | Arm E (Ixazomib Citrate, Cyclophosphamide, Daratumumab) (N=24)
Anemia (Blood and lymphatic system disorders) | 9 (22) | 6 (59) | 4 (12) | 16 (237) | 22 (291)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (122) | 19 (100) | 21 (134) | 24 (147) | 18 (61)
Diarrhea (Gastrointestinal disorders) | 26 (234) | 24 (174) | 25 (113) | 29 (208) | 17 (146)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (5)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 28 (144) | 19 (71) | 23 (103) | 28 (124) | 16 (103)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (37) | 9 (15) | 11 (22) | 11 (19) | 7 (23)
Edema limbs (General disorders) | 13 (114) | 14 (120) | 14 (92) | 21 (145) | 17 (224)
Fatigue (General disorders) | 29 (430) | 33 (441) | 29 (355) | 34 (514) | 22 (421)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 3 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 11 (130) | 13 (59) | 9 (15) | 19 (127) | 13 (59)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 10 (181) | 8 (47) | 11 (55) | 25 (394) | 22 (307)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 15 (52) | 15 (31) | 17 (59) | 23 (135) | 8 (44)
Platelet count decreased (Investigations) | 27 (244) | 26 (148) | 28 (144) | 26 (371) | 17 (69)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 5 (24) | 7 (13) | 9 (24) | 9 (48) | 7 (24)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (13) | 2 (8) | 2 (7) | 5 (57) | 6 (57)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (18)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (5) | 1 (2) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 11 (36) | 8 (48) | 5 (59) | 13 (89) | 4 (11)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (5) | 0 (0) | 1 (6) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (5)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 11 (30) | 7 (93) | 8 (50) | 8 (34) | 8 (117)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (346) | 31 (345) | 27 (384) | 25 (439) | 20 (363)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (8) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (20) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (13) | 2 (12) | 5 (68) | 9 (29) | 5 (22)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (30) | 13 (53) | 11 (31) | 8 (32) | 10 (23)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT01415882/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT01415882/ICF_001.pdf